CLINICAL TRIAL: NCT05713123
Title: Comparison of a 3D Recording in a VERITON-CT™ Camera to the Anger Camera Procedure in Patients Treated by Iodine 131 for a Thyroid Cancer
Brief Title: Comparison of Record in VERITON Camera to the Anger Camera Procedure in Patients Treated by 131-iodine
Acronym: VERICATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Elodie CHEVALIER, Principal investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021PI234
Record Dates: First submitted 2022-12-06; First posted 2023-02-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Device
Keywords: Iodine 131; Thyroid cancer; Camera CZT (cadmium-Zinc-Tellurid)
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients received Iode 131 for thyroid cancer and 72 hours after taking iodine capsule,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Person suffering from thyroid cancer and treated by iodine 131 (1100 MBq or 3700 MBq) (Experimental): The study will be offered to patients suffering from thyroid cancer and treated by iodine 131 (1100 MBq or 3700 MBq). When they come in nuclear medicine to have the iodine scan in Anger's camera, if they signed the consent, they will the SPECT/CT whole body in VERITON-CT camera
  Interventions: Other: A SPECT-CT whole body is added in VERITON-CT camera

INTERVENTIONS:
Other: A SPECT-CT whole body is added in VERITON-CT camera — A SPECT-CT whole body in VERITON-CT camera is added after the conventional procedure recorded in Anger camera

SUMMARY:
The aim of this study is to show that the SPECT/CT whole body recording procedure lasting less than or equal to 30 minutes in a VERITON-CT™ camera, can be substituted for the classic procedure, giving at least equivalent information in searches for primary or metastatic neoplastic lesions.

DETAILED DESCRIPTION:
Patients with thyroid cancer treated with iodine 131 will receive an iodine 131 activity of between 1100 and 3700 MBq delivered as a capsule orally to eliminate the remaining thyroid tissue. Hormone replacement therapy (HRT) is then started to correct the hypothyroidism.

3 days later, a 2D whole body recording will be associated with complementary Single Photonic Emission Computed Tomography CT scans (SPECT/CT). It enables visualising the fixation of iodine 131, provides information on the thyroid remnants left in place during surgical thyroidectomy and to carry out an extension assessment by visualizing the possible presence of metastases fixing iodine at the level of the regional lymph nodes or many distant sites, in particular, lung and bone.

In VERICATH study, the hypothesis is that this classic procedure could be advantageously replaced by a single full-body SPECT/CT recording of a limited duration (≤ 30 minutes), obtained with a camera state-of-the-art semiconductor device called the VERITON-CT™ (Spectrum Dynamics Medical) camera.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18, who have understood and signed the informed consent form.
2. Person suffering from thyroid cancer and for whom the multidisciplinary meeting has validated a treatment by iodine 131 (1100 MBq or 3700 MBq).
3. Person with no contraindication to carrying out the examination.
4. Person affiliated to a social security scheme.

Exclusion Criteria:

1. Person with a known allergy to one of the components of the radiopharmaceutical (Iodine 131 capsule).
2. Pregnant woman or woman of childbearing age and without suitable contraceptive means, or breastfeeding mother.
3. Person whose medical condition is unstable and/or unable to remain still in the supine position during recordings.
4. Person deprived of liberty by a judicial or administrative decision.
5. Person of full age subject to a measure of legal protection (guardianship, curators, safeguard of justice).
6. Adult person unable to express his consent and who is not the subject of a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2025-04-26 (Estimated)

PRIMARY OUTCOMES:
Compare post-therapy imaging performed with the two procedures | 18 months
  Type of lesions
  * Lesions
  * The nature of the lesion(s): thyroid residue and/or lymph node lesion and/or metastases (distant lesions).
  * Number of lesions in conventional camera and in VERITON-CT™ camera.

SECONDARY OUTCOMES:
Compare the two procedures in terms of cancer status result. | 18 months
  Status of cancer
Determine the feasibility of a 3D quantification of the fixation of thyroid residues in a VERITON-CT™ camera | 18 months
  Measurement of absolute quantification with the 2 procedures
Evaluate the two exams in terms of ergonomics for technologists | 18 months
  Likert scale results

CONTACTS AND LOCATIONS:
Overall Officials: Elodie CHEVALIER, MD, Principal Investigator — CHRU Nancy
Locations (1):
- Chru Nancy Brabois, Vandœuvre-lès-Nancy, France